CLINICAL TRIAL: NCT05439148
Title: A Phase I, Open-label, Single- and Multi-Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacological Effect of OPC-61815 in Healthy Chinese Male Subjects
Brief Title: OPC-61815 in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 263-403-00011
Record Dates: First submitted 2022-04-18; First posted 2022-06-30 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-02

CONDITIONS: Healthy Adult Male

STUDY DESIGN:
Intervention Model Description: 8 mg and 16 mg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OPC-61815 (Experimental): Intravenous administration of OPC-61815 at 8 mg or 16 mg. 8mg group will be intravenously administered only on D1, once a day. 16mg group will be intravenously administered on D1，D3-D9, once a day
  Interventions: Drug: OPC-61815 injection

INTERVENTIONS:
Drug: OPC-61815 injection — Intravenous administration of OPC-61815 at 8 mg or 16 mg. 8mg group will be intravenously administered only on D1, once a day. 16mg group will be intravenously administered on D1，D3-D9, once a day.

SUMMARY:
To evaluate the pharmacokinetic (PK) characteristics and pharmacological effect of OPC-61815 in healthy Chinese Male subjects

DETAILED DESCRIPTION:
To evaluate the pharmacokinetic (PK) characteristics of single and multiple intravenous administration of OPC-61815 in healthy Chinese subjects.

To evaluate the safety of single and multiple intravenous administration of OPC-61815 in healthy Chinese subjects.

To evaluate the pharmacological effect of single and multiple intravenous administration of OPC-61815 in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18-45 years (including the cutoff values, subject to the time of signing the Informed Consent Form (ICF));
* Body mass index (BMI) of 19-26 kg/m2 (including the cutoff values), with a body weight of not less than 50 kg for male subjects;

Exclusion Criteria:

* Those whose the sitting pulse is lower than 50 beats/min or higher than 100 beats/min after resting for over 3 minutes.
* Those whose sitting SBP is lower than 90 mmHg or higher than 140 mmHg, or DBP is lower than 50 mmHg or higher than 90 mmHg after resting for over 3 minutes.
* Various micturition disorders (pollakiuria or dysuria, etc.).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic (PK) characteristics：Tmax | before dosing and after the start of dosing on Day1 and Day9(16mg group only); 16mg group also need collect on Day7 and Day8
  Pharmacokinetic parameters of OPC-61815 free form and metabolites tolvaptan, DM4103 and DM4107 in plasma after intravenous administration of OPC-61815
To evaluate the pharmacokinetic (PK) characteristics：Cmax | before dosing and after the start of dosing on Day1 and Day9(16mg group only); 16mg group also need collect on Day7 and Day8
  Pharmacokinetic parameters of OPC-61815 free form and metabolites tolvaptan, DM4103 and DM4107 in plasma after intravenous administration of OPC-61815
To evaluate the pharmacokinetic (PK) characteristics：AUC0-t, AUC0-inf, AUC0-24h | before dosing and after the start of dosing on Day1 and Day9(16mg group only); 16mg group also need collect on Day7 and Day8
  Pharmacokinetic parameters of OPC-61815 free form and metabolites tolvaptan, DM4103 and DM4107 in plasma after intravenous administration of OPC-61815
To evaluate the pharmacokinetic (PK) characteristics：t1/2 | before dosing and after the start of dosing on Day1 and Day9(16mg group only); 16mg group also need collect on Day7 and Day8
  Pharmacokinetic parameters of OPC-61815 free form and metabolites tolvaptan, DM4103 and DM4107 in plasma after intravenous administration of OPC-61815
To evaluate the pharmacokinetic (PK) characteristics：λz | before dosing and after the start of dosing on Day1 and Day9(16mg group only); 16mg group also need collect on Day7 and Day8
  Pharmacokinetic parameters of OPC-61815 free form and metabolites tolvaptan, DM4103 and DM4107 in plasma after intravenous administration of OPC-61815
To evaluate the pharmacokinetic (PK) characteristics：Rac(Cmax) | before dosing and after the start of dosing on Day1 and Day9(16mg group only); 16mg group also need collect on Day7 and Day8
  Pharmacokinetic parameters of OPC-61815 free form and metabolites tolvaptan, DM4103 and DM4107 in plasma after intravenous administration of OPC-61815
To evaluate the pharmacokinetic (PK) characteristics：Rac(AUC0-24h) | before dosing and after the start of dosing on Day1 and Day9(16mg group only); 16mg group also need collect on Day7 and Day8
  Pharmacokinetic parameters of OPC-61815 free form and metabolites tolvaptan, DM4103 and DM4107 in plasma after intravenous administration of OPC-61815
To evaluate the pharmacokinetic (PK) characteristics：CL (OPC-61815 free form only) | before dosing and after the start of dosing on Day1 and Day9(16mg group only); 16mg group also need collect on Day7 and Day8
  Pharmacokinetic parameters of OPC-61815 free form in plasma after intravenous administration of OPC-61815
To evaluate the pharmacokinetic (PK) characteristics：Vz (OPC-61815 free form only) | before dosing and after the start of dosing on Day1 and Day9(16mg group only); 16mg group also need collect on Day7 and Day8
  Pharmacokinetic parameters of OPC-61815 free form in plasma after intravenous administration of OPC-61815

SECONDARY OUTCOMES:
To evaluate the safety of single and multiple intravenous administration：laboratory tests | from screening period to follow up period,assessed up to 16 Days.
  laboratory tests assessment variables include blood routine, blood biochemistry and urine routine.
To evaluate the safety of single and multiple intravenous administration：adverse events | from screening period to follow up period,assessed up to 16 Days.
  adverse events start date, end date , seriousness, severity, relationship to trial treatment (IMP causality), action taken with trial treatment, and outcome will be collect

CONTACTS AND LOCATIONS:
Overall Officials: Hongyun Wang, Principal Investigator — Peking Union Medical College Hospital; Hongzhong Liu, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Clinical Pharmacology Research Center, Peking Union Medical College Hospital, Beijing, China